CLINICAL TRIAL: NCT06766344
Title: Examınatıon of Sports Injury Anxıety Level and Sports Injury Preventıon Awareness of Unıversıty Students Partıcıpatıng in Sports
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Betul Ergun, Lecturer, Inonu University
Other Study IDs: SPORTS INJURY
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Sport Injuries
Keywords: Awareness; Sport; Injury; Students
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Faculty of Sports Sciences
- Faculty of Health Sciences
- Faculty of Medicine

SUMMARY:
This study aimed to evaluate the concerns of university students who are involved in sports on more than one subject related to sports injuries (anxiety of losing ability, anxiety of suffering, anxiety of losing social support, etc.). In addition, in this study, the awareness of protection from sports injuries was evaluated in order to minimize sports injuries and create awareness of injury prevention, based on the idea that the athlete will be injured less with less anxiety in sports life.

DETAILED DESCRIPTION:
Regardless of the sport branch, athletes are likely to encounter many injury stories during their active sports life. Stories of sports injuries cause anxiety in athletes. Therefore, sports injury prevention awareness is important. This study aimed to evaluate and compare the anxiety about sports injuries and sports injury prevention awareness of university students studying in different faculties and practicing regular sports. Personal Information Form, Sports Injury Anxiety Scale (SIAS) and Sports Injury Prevention Awareness Scale (SIPAS) were used. There was no difference between university students from three different faculties who participated in sports in terms of the total scores of the SIAS and SIPAS (p>0.05). It was determined that there was a significant difference between the students from three faculties in terms of the Anxiety of Losing Ability (ALA) parameter, which is one of the subscales of the SIAS (p<0.05). In pairwise comparisons between the groups, a significant difference was found between the students of health sciences and medical faculties in the subscale of the SIAS-ALA (p=0.001). University students who participated in sports from all three faculties included in the study had normal levels of anxiety about sports injuries and high levels of sports injury awareness. High sports injury awareness of students participating in sports may be an important factor for injury prevention. Low levels of anxiety may also be associated with high levels of awareness.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* To be a student in one of the Faculties of Sports Sciences, Health Sciences, Engineering and Medicine
* Participating in a regular sport branch

Exclusion Criteria:

* - Being diagnosed with a chronic disease or regular medication use
* Not being a student in one of the Faculties of Sports Sciences, Health Sciences, Engineering and Medicine
* Voluntary separation from employment
* Failure to complete the questionnaires to be applied within the scope of the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The study was conducted on university students participating in various sports branches, especially volleyball, basketball, soccer, swimming, fitness, pilates, walking. A total of 126 volunteer university students who regularly participated in sports were included in the study. Those with a history of chronic disease or regular medication use were excluded from the study, and those who did not complete the survey questions required for the study were excluded from the study.
  In the power analysis performed to determine the sample size, the type I error was 0.05 and the type II error was 0.2. The power was set at 0.8. Power analysis was performed using the G-Power 3.1.7 package (Heinrich-Heine-University, Düsseldorf, Germany). The minimum number of subjects to be included in the study in each group was determined as 18 in order to find a mean difference of 3 units significant according to the Sports Injury Anxiety Scale sub-dimension score.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
assessment of sports injury anxiety among students | Day 1 (when students first arrive)
  Examınatıon of Sports Injury Anxıety Level of Unıversıty Students Partıcıpatıng in Sports. Their thoughts and anxiety levels about sports injury were evaluated with the 'Sports Injury Anxiety Scale', whose Turkish validity and reliability study was conducted by Caz et al. (2019). The scale consists of 19 items in total. It consists of sub-dimensions such as loss of ability, suffering, perceived weakness, loss of social support, disappointment, and anxiety of re-injury. A 5-point Likert scale was used in the evaluation. The survey questions were answered as "1=Strongly Disagree" and "5=Strongly Agree". The lowest score that can be obtained from the scale is 19 and the highest score is 95.

SECONDARY OUTCOMES:
evaluation of students' awareness of protection from sports injuries | Day 1 (when students first arrive)
  Examınatıon of Sports Injury Preventıon Awareness of Unıversıty Students Partıcıpatıng in Sports. The knowledge levels of the participants about sports injuries and protection from sports injuries were evaluated with the Sports Injury Protection Awareness Scale developed by Ercan and Önal in 2021. It consists of 18 items in total. Sub-dimensions in the scale; personal health status is examined with items 1-4, environmental factors and equipment with items 5-9, exercise session with items 10-14, and exercise program with items 15-18. A 5-point Likert scale was used in the evaluation. Survey questions were answered as "1=Strongly Disagree", "2=Disagree", "3=Undecided", "4=Agree", "5=Strongly Agree".

CONTACTS AND LOCATIONS:
Locations (1):
- Inönü University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No